CLINICAL TRIAL: NCT00903955
Title: SCCOR in Host Factors in Chronic Lung Disease
Brief Title: Mucus Dehydration and Evolution of Chronic Obstructive Pulmonary Disease (COPD) Lung Disease
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Richard C Boucher, MD, Director of Cystic Fibrosis Center, University of North Carolina, Chapel Hill
Other Study IDs: 05-2876; 5P50HL084934-02 (NIH)
Record Dates: First submitted 2009-05-17; First posted 2009-05-19 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Chronic Obstructive Pulmonary Disease; Chronic Bronchitis
Keywords: Mucus; COPD; Chronic Bronchitis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic | interventions — Saline Solution, Hypertonic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Chronic Obstructive Pulmonary Disease: Subjects diagnosed with COPD are classified according to standards set forth by the Global Initiative on Obstructive Lung Disease. This study recruits subjects in each of three GOLD categories.
  Interventions: Other: 7% hypertonic saline

INTERVENTIONS:
Other: 7% hypertonic saline — Administered via jet nebulizer to subjects in specific aim 3

SUMMARY:
The purpose of this research is to understand the properties of mucus in persons with COPD, specifically Chronic Bronchitis. We hypothesize that those with Chronic Bronchitis have dehydrated mucus, and thus have a harder time coughing it out of their lungs. This leads to a greater vulnerability for lung infection, inflammation and airflow obstruction. Ultimately, our goal is to understand how mucus dehydration contributes to the progression of COPD/Chronic Bronchitis so that better therapies and interventions can be developed for future generations.

DETAILED DESCRIPTION:
Specific Aim I directly tests the hypothesis that mucus clearance is impaired due to mucus dehydration. It measures 1) COPD Mucociliary and Cough Clearance 2) mucus hydration 3) the concentrations of the dominant regulators of airway hydration and 4) the consequences of mucus dehydration on mucus biophysical properties and bacterial infection.

Specific Aim II tests the hypothesis that COPD acute exacerbations are associated with failures of mucus clearance. Measurements will be similar to that of Specific Aim I, but conducted during periods of baseline health, acute exacerbation and recovery.

Specific Aim III tests whether airway surface hydration with 7% Hypertonic Saline will restore clearance in the basal state and during a COPD acute exacerbation. COPD subjects will be exposed to inhaled Hypertonic Saline during periods of baseline health and acute exacerbation. Acute efficacy via measures of mucus clearance and spirometry will studied.

ELIGIBILITY:
Inclusion Criteria:

* history of COPD/chronic bronchitis defined as having a productive cough for three months of the year for at least two successive years
* greater than or equal to a 10 pack year cigarette smoking history
* ability to perform spirometry

Exclusion Criteria:

* unstable lung disease
* allergy to study medications
* radiation exposure within past year exceeding Federal Regulation Limits

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community members with a history of cigarette smoking and COPD/chronic bronchitis.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2006-09; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Mucociliary clearance of inhaled tc99m | 24 hours

SECONDARY OUTCOMES:
Identification of bacterial and viral communities in mucus samples; analysis of biochemical and biophysical properties of mucus | March 2012

CONTACTS AND LOCATIONS:
Overall Officials: Richard Boucher, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina Chapel Hill, Chapel Hill, North Carolina, United States